CLINICAL TRIAL: NCT06466538
Title: Effectiveness of Boswellia as Intracanal Medication on Infectious/Inflammatory Contents in Teeth With Apical Periodontitis
Brief Title: Investigate"Clinically" the Effectiveness of Boswellia Based Intracanal Medication Compared to Calcium Hydroxide Ca(OH)2 and Ledermix on the Levels of Bacteria and Inflammatory Cytokines in Root Canals and Periradicular Tissues of Teeth With Apical Periodontitis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Root Canal Medicament
Record Dates: First submitted 2024-06-08; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases | interventions — Calcium Hydroxide; Frankincense

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calcium Hydroxide (Active Comparator): intracanal medicament
  Interventions: Drug: Calcium hydroxide
- Leddermix (Active Comparator): intracanal medicament
  Interventions: Drug: Leddermix
- Boswellia (Active Comparator): intracanal medicament
  Interventions: Drug: Boswellia

INTERVENTIONS:
Drug: Calcium hydroxide — intracanal medicament
  Arms: Calcium Hydroxide
Drug: Leddermix — Leddermix
  Arms: Leddermix
Drug: Boswellia — Boswellia
  Arms: Boswellia

SUMMARY:
The objective of this study is to investigate "clinically" the effectiveness of Boswellia based intracanal medication compared to the commonly used intracanal medicaments (calcium hydroxide Ca(OH)2 and Ledermix) on the levels of bacteria and inflammatory cytokines in root canals and periradicular tissues of teeth with apical periodontitis.

DETAILED DESCRIPTION:
Apical periodontitis is an inflammatory disorder of the periradicular tissue caused by bacterial infection of endodontic origin, which is characterized by periapical bone resorption. Primary endodontic disease has a polymicrobial etiology, with predominance of Gram-negative anaerobic bacteria. This species presents lipopolysaccharides (LPSs), one of the most important inflammatory molecules present in the outer layer of its membrane, which can be released during multiplication or bacterial death, thus continuously stimulating the surrounding tissues even at low levels.

Endotoxins have been detected in 100% of the primarily infected root canals, with high levels being related to more severe inflammatory response in periapical tissues. When bacteria and their toxins (e.g., LPS) present in the root canal infection egress into the periapical tissues via apical foramen, they activate immune response locally, culminating in a very complex inflammatory disorder involving a variety of inflammatory cells as well as different proinflammatory cytokines. IL-1β, TNF-α, and PGE2 have been detected in periapical tissues, being considered important inflammatory biomarkers in the apical disease. Since bacteria and their by-products are one of the main causes of apical periodontitis, special emphasis is given to the search for an optimal root canal disinfection protocol.

Although instrumentation may be assumed to be of greater importance in the clinical practice, the use of intracanal medication has been proven to optimize the root canal disinfection. For this reason, a wide variety of intracanal medications have been proposed. Calcium hydroxide [Ca(OH)2] is the most commonly used intracanal medication. Lately, chlorhexidine (CHX) has emerged as a potential intracanal medication and suggested to be used alone or combined with Ca(OH)2 in a paste. Although studies have investigated the antibacterial property of Ca(OH)2, including CHX associations, the effects on immune periapical response is incipient.

Another effective intracanal medication is Ledermix which contains 1% triamcinolone (TAA) and 3% demeclocycline (DOC). This formulation was first recommended for use in endodontics. The use of Ledermix appear to be more likely related to the anti-inflammatory effects of corticosteroid rather than its antibacterial effect .The antibiotic component does not appear to be ideal, and the use of other antibiotics may help to improve the antimicrobial effects of Ledermix.

Because root canal medicaments can come in contact with periapical tissue, in addition to having good antibacterial ability, they must also be biocompatible. In selecting root canal medicaments, it is necessary to consider their therapeutic benefits against their potential cytotoxic effects. Ideal root canal medicaments should have strong antibacterial properties and minimal cytotoxic effect on the host tissues. Herbs have been used in clinical medicine for thousands of years. However, it is only in recent times that researchers have been able to employ scientific methods to prove the efficacy of many of these herbs and to provide a better understanding of their mechanisms of action (Graf 2000).

Ayurveda (Indian traditional medicine practice) used Boswellia for the treatment of gastrointestinal diseases such as diarrhea, constipation, flatulence and vomiting. It was also stated that the extract is useful in the treatment for diabetic patients and also for respiratory complications including cough, cold, hoarseness, bronchitis, asthma and dyspnea.

So based on the above mentioned data, it is believed to be of interest to investigate clinically the use of Boswellia as an intracanal medication.

ELIGIBILITY:
Inclusion Criteria:

* Single-rooted with pulp necrosis and apical periodontitis.
* The age range from 20 to 60 years

Exclusion Criteria:

* Receiving antibiotic treatment within the preceding 3 months.
* Reporting systemic disease.
* Teeth that could not be isolated with rubber dam.
* Teeth with periodontal pockets deeper than 3 mm.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Microbiological culture (manual counting to bacterial cells) | up to 8 months
  Bacterial counting after culturing of bacteria

SECONDARY OUTCOMES:
ELISA test to measure levels of Inflammatory cytokines (tumor necrotizing factor, prostaglandin E2, Interleukin 1B) | 30 weeks
  ELISA test to measure levels of Inflammatory cytokines (tumor necrotizing factor, prostaglandin E2, Interleukin 1B)

CONTACTS AND LOCATIONS:
Overall Officials: Amany Badr, Professor, Study Chair — Mansoura University; Youssry RM Elhawary, Professor, Study Director — Mansoura University
Locations (1):
- May Abuzoor, Al Mansurah, Egypt

REFERENCES:
- [Background] Khosravi Samani M, Mahmoodian H, Moghadamnia A, Poorsattar Bejeh Mir A, Chitsazan M. The effect of Frankincense in the treatment of moderate plaque-induced gingivitis: a double blinded randomized clinical trial. Daru. 2011;19(4):288-94. PMID 22615671
- [Background] Raja AF, Ali F, Khan IA, Shawl AS, Arora DS, Shah BA, Taneja SC. Antistaphylococcal and biofilm inhibitory activities of acetyl-11-keto-beta-boswellic acid from Boswellia serrata. BMC Microbiol. 2011 Mar 16;11:54. doi: 10.1186/1471-2180-11-54. PMID 21406118